CLINICAL TRIAL: NCT00213460
Title: Small Bowel Motor Impairment in Scleroderma: Results of a Prospective 5-year Manometric Follow-up
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2000/103/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Small bowel involvement is still recognized to be associated with great morbidity and mortality in SSc patients, leading particularly to malabsorption and intestinal pseudo-obstruction. Intestinal disorders directly related to SSc have, in fact, been reported to be one of the most common causes of death.

In a previous prospective study, we have demonstrated the high prevalence of small intestinal involvement in SSc patients, using upper intestinal manometry; in turn, 88% of our SSc patients had upper intestinal motor disturbances. However, to date, no authors have yet analyzed the course of upper intestinal motor dysfunction in SSc.

The aims of this study were therefore to assess the 5-year course of small bowel motor disorders, using manometry in patients with systemic sclerosis (SSc), and to investigate for an association between upper intestinal motor dysfunction outcome and other clinical manifestations of SSc.

ELIGIBILITY:
Inclusion Criteria:

* patients with systemic sclerosis, who had an upper intestinal tract manometry 5 years before, with:

  * age over 18 years
  * written informed consent

Exclusion Criteria:

* pregant women
* patients with psychiatric conditions
* unwritten informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-08; Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle MARIE, MD, PhD, Principal Investigator — CHU Rouen
Locations (1):
- CHU Rouen, Rouen, Rouen Cedex, France